CLINICAL TRIAL: NCT05898490
Title: The Effect of Animation Therapy on Time Perception in Primary School Children: A Randomized Controlled Study
Brief Title: The Effect of Animation Therapy on Time Perception in Primary School Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ozgun Belen, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03/06
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Time Perception Altered
Keywords: time perception; animation therapy; occupational therapy; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation Therapy Group (Experimental): 10 sessions of Animation Therapy (2 session/week)
  Interventions: Behavioral: Animation Therapy
- Control Froup (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Animation Therapy — The process of shooting a stop-motion animation film, is designed according to the interests and leading of the participant.
  Arms: Animation Therapy Group

SUMMARY:
The aim of the study is to determine the effects of animation therapy on time perception and daily activity routine performances of primary school children.

DETAILED DESCRIPTION:
Time is a process that forms the basis of executive functions used to reveal adaptive behavior and motor performance. However, the way we perceive time can be changed by different factors. This may reveal changes in executive functions such as decision making, behavioral inhibition, planning, and accordingly, in the performance levels and daily routines of daily living activities. Animation therapy is the therapeutic use of the process of shooting a stop-motion animation film. It creates a "flow" effect by nature. The concept of flow includes the loss of the sense of time. In this study, it is aimed to examine whether animation therapy has an effect on the perception of time and daily activity routines in primary school children.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7-10
* Absence of any orthopedic, neurodevelopmental, and psychiatric problems/diagnosis
* Continuing formal education
* Voluntarily agreeing to participate in the research

Exclusion Criteria:

* Receiving orthopedic, neurodevelopmental and psychiatric diagnosis during the study period
* To be absent from the study process or to quit the process
* Not participating in the first and last evaluations
* Voluntary refusal to participate or continue with the research

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Time Discrimination Task | Baseline, preintervention
  Time Discrimination Task is based on the individual's perception of the time difference of two different gaps between two pairs of sequentially given stimuli. Generally, the person is asked to indicate which pair is longer or shorter between two pairs of stimuli of certain lengths, which are given visually and/or audibly. Leveling is performed with the UDTR (Up-Down Transformed-Response) adaptive procedure method to progress the test and determine the participant's discrimination threshold.
Time Discrimination Task | Immediately after the intervention
  Time Discrimination Task is based on the individual's perception of the time difference of two different gaps between two pairs of sequentially given stimuli. Generally, the person is asked to indicate which pair is longer or shorter between two pairs of stimuli of certain lengths, which are given visually and/or audibly. Leveling is performed with the UDTR (Up-Down Transformed-Response) adaptive procedure method to progress the test and determine the participant's discrimination threshold.
Time Reproduction Task | Baseline, preintervention
  In Time Reproduction Task, the participants are asked to produce a stimulus similar to the duration of the stimulus presented to them at certain durations. In our study, visual and auditory stimuli of 200ms, 500ms and 800ms will be presented to the person in the time reproduction task, as in the time discrimination task. These stimuli will be presented in a completely random order, not in a specific order, and each stimulus will be presented 10 times, with a total of 30 consecutive stimuli. A gap of 2000 ms will be left between both stimuli to allow enough time for the person to reproduce the stimulus. The ratio of the absolute value of the difference between the participant's reproduced time and the target time to the target time will be calculated.
Time Reproduction Task | Immediately after the intervention
  In Time Reproduction Task, the participants are asked to produce a stimulus similar to the duration of the stimulus presented to them at certain durations. In our study, visual and auditory stimuli of 200ms, 500ms and 800ms will be presented to the person in the time reproduction task, as in the time discrimination task. These stimuli will be presented in a completely random order, not in a specific order, and each stimulus will be presented 10 times, with a total of 30 consecutive stimuli. A gap of 2000 ms will be left between both stimuli to allow enough time for the person to reproduce the stimulus. The ratio of the absolute value of the difference between the participant's reproduced time and the target time to the target time will be calculated.
Executive Functions and Occupational Routines Score | Baseline, preintervention
  This scale evaluates children's performance in daily activity routines, was developed by Fisch and Rosenblum in 2014. This scale evaluates the daily routines and executive functions of children aged 6-12 years, according to the opinion of their parents/caregivers. It consists of 3 sub-dimensions: Morning and Evening Routines (16 items), Game and Leisure Routines (7 items), and Social Routines (7 items). It is in the form of a five-point Likert scale and each item can be scored between 1 (never) and 5 (always). A high score indicates that the child's performance is high. The scale, which consists of 30 items in total, can be completed in approximately 15 minutes.
Executive Functions and Occupational Routines Score | Immediately after the intervention
  This scale evaluates children's performance in daily activity routines, was developed by Fisch and Rosenblum in 2014. This scale evaluates the daily routines and executive functions of children aged 6-12 years, according to the opinion of their parents/caregivers. It consists of 3 sub-dimensions: Morning and Evening Routines (16 items), Game and Leisure Routines (7 items), and Social Routines (7 items). It is in the form of a five-point Likert scale and each item can be scored between 1 (never) and 5 (always). A high score indicates that the child's performance is high. The scale, which consists of 30 items in total, can be completed in approximately 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Prof., Study Director — Hacettepe University; Özgün Belen, MSc, Principal Investigator — Kütahya Health Sciences University
Locations (1):
- Özel Yaşam Köyü İlkokulu, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No